CLINICAL TRIAL: NCT03097081
Title: Orthosis Versus no Orthosis After Dorsally Fixated Traumatic Thoracolumbar Fractures
Brief Title: ORthosis vs No Orthosis After Surgically Treated Traumatic Thoracolumbar Fractures
Acronym: ORNOT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, AJ Smits, MD, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ORNOT-trial
Record Dates: First submitted 2017-03-20; First posted 2017-03-31 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Spine Fracture; Orthosis; Traumatic Fracture; Posterior Fixation
MeSH Terms: conditions — Spinal Fractures | interventions — Orthotic Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No orthosis (Experimental): The intervention consists of a deviation of the standard protocol; patients post-operatively do not receive an orthosis.
  Interventions: Other: No orthosis
- Orthosis (Active Comparator): As in correspondence with local and international guidelines, patients receive an orthosis as standard post-operative care. This is considered the control group.
  Interventions: Device: Orthosis

INTERVENTIONS:
Other: No orthosis — The intervention consists of a deviation of the standard protocol; patients do not receive a post-operative orthosis
  Arms: No orthosis
Device: Orthosis — Patients receive post-operative care following the standard protocol and wear an orthosis for 10-12 weeks.
  Arms: Orthosis

SUMMARY:
Rationale: There is no evidence in the current literature regarding the additional value of an orthosis after surgically treated thoracolumbar spine fractures.

Objective: To assess whether an orthosis provides additional pain relief compared to no orthosis after posteriorly fixated thoracolumbar spine fractures. Primary outcome is difference in pain at six weeks post-operatively. Secondary objectives are pain at other moments, pain medication used, pain related disability, quality of life, long-term kyphosis, possible complications, hospital stay, return to work and subjective feeling on benefit or disadvantage from the orthosis.

Study design: Randomized controlled intervention study, non-inferiority trial.

Study population: Dutch speaking patients presented at the VU university medical centre, 18 - 65 years old with a traumatic thoracolumbar spine fracture from Th7 - L4 surgically treated by posterior fixation.

Intervention: One group receives standard care and wears an orthosis after surgery for 12 weeks, to use when in vertical position. The intervention group does not wear an orthosis after surgery.

Main study parameters/endpoints: Main study outcome is the difference in pain noted on the NRS-score at six weeks, ≥ 2 (SD 2,5) change corresponds with a clinically significant change in pain score.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The current guideline for postoperative care regarding dorsal stabilization of spine fractures recommends the use of a post-operative orthosis. While patients generally receive an orthosis for 12 weeks, individual surgeon's believes sometimes gives reason to deviate from this guideline. This is founded by literature that increasingly questions the use of orthoses in the conservative treatment of spine fractures. With the fracture operatively stabilized, the orthosis mainly provides support of gesture and thereby potentially results in pain relief and confidence for patients. On the other hand some patients have a hard time weaning from the orthosis or report discomfort due to the device and prefer not to use it. With subjects being randomized between the use of an orthosis or no orthosis there is no additional risk. This is in part because it is hypothesized that there is no difference in postoperative pain and there might be a lower risk of complications related to the orthosis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 65 years
* Traumatic thoracolumbar spine fracture from thoracic 7 - lumbar 4
* AO fracture types A-C
* Undergoing surgical dorsal fixation for fracture

Exclusion Criteria:

* Inadequate knowledge of Dutch language or to fill in questionnaire
* Complete or partial spinal cord injury (ASIA A to D)
* (Additional) anterior surgical stabilization
* Thoracolumbar fracture of other aetiology than traumatic, e.g. pathologic, infectious
* Not able to walk before fracturing vertebra
* Unable to come to the outpatient clinic (e.g. residing outside the Netherlands)
* Injury Severity Score (ISS) ≥ 16
* Brain injury with Abbreviated Injury Score (AIS) ≥ 4
* Solitary Lumbar 5 fracture
* Inability to wear an orthosis, most probable reasons:

  * BMI > 35
  * Thoraco-abdominal wounds (through trauma or secondary from surgery) on places at which the orthosis contacts the body so aggravation of pain or chances of infection increase significantly.

    12 of 27
  * Pre-existing spine deformities (scoliosis or very severe kyphosis/lordosis) which impair the use of the orthosis or aggravate pain.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2016-11; Primary Completion 2025-01 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Pain (NRS) | 6 weeks

SECONDARY OUTCOMES:
Pain (NRS) | Post-operative, 2 & 12 weeks
Quality of life (EQ-5D) | Post-operative, 12 weeks & 6, 12 months
Back pain related function (ODI) | Post-operative, 2, 6, 12 weeks & 6, 12 months
Kyphosis (Cobb-angle) | Pre-operative, post-operative, 6, 12 weeks & 6, 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- VU University medical center, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Derived] Smits AJ, Deunk J, Stadhouder A, Altena MC, Kempen DHR, Bloemers FW. Is postoperative bracing after pedicle screw fixation of spine fractures necessary? Study protocol of the ORNOT study: a randomised controlled multicentre trial. BMJ Open. 2018 Jan 13;8(1):e019596. doi: 10.1136/bmjopen-2017-019596. PMID 29331975